CLINICAL TRIAL: NCT02099539
Title: A Phase I/II Study of N-803 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: QUILT-3.005: A Study of N-803 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: Altor BioScience (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-803-02-13; CA167925 (Other: NIH)
Record Dates: First submitted 2014-02-26; First posted 2014-03-31 (Estimated); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2018-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: absolute lymphocyte count; antitumor; cancer; immunotherapy; immunochemotherapy; interleukin-15; multiple myeloma; NK cell; refractory; relapsed; T cell; white blood cell count
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Neoplasms | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1: N-803 - IV 1 ug/kg (Experimental)
  Interventions: Biological: N-803
- Cohort 2: N-803 - IV 3 ug/kg (Experimental)
  Interventions: Biological: N-803
- Cohort 3: N-803 - IV 6 ug/kg (Experimental)
  Interventions: Biological: N-803
- Cohort 4: N-803 - IV 10 ug/kg (Experimental)
  Interventions: Biological: N-803
- Cohort 5: N-803 - SQ 10 ug/kg (Experimental)
  Interventions: Biological: N-803
- Cohort 6: N-803 - SQ 15 ug/kg (Experimental)
  Interventions: Biological: N-803

INTERVENTIONS:
Biological: N-803 — Intravenous infusion for cohort 1, 2, 3 and 4; subcutaneous injection for cohort 5, 6 and 7; two 6-week treatment cycles: ALT-803 on Day 1, 8, 15, 22; stable or benefitting patients may receive up to two additional 6-week cycles

SUMMARY:
This is a Phase I/II, open-label, multi-center, competitive enrollment and dose escalation study of N-803 in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, determine the Maximum Tolerated Dose (MTD) or the Minimum Efficacious Dose (MED) and characterize the immunogenicity and pharmacokinetic profile of N-803 in treated patients. The effect of N-803 on the peripheral absolute lymphocyte counts and white blood cell counts, the number and phenotype of peripheral blood T (total and subsets) and NK cells will be evaluated. The anti-tumor responses of N-803 will also be assessed in this trial.

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARACTERISTICS:

* Confirmed diagnosis of relapsed/refractory multiple myeloma after treatment with at least two different previous regimens.

  * Refractory disease is defined as progressive disease while on therapy or progression within 60 days of therapy.
  * Progressive disease is defined by a 25% increase from the lowest response value in specified tests.
* Measurable disease as defined by at least one of the following:

  * Serum M-protein ≥ 1g/dL (for IgG, IgM) or 0.5 g/dL (for IgA)
  * Urine M-protein ≥ 200mg/24hours
  * Serum free light chains ≥ 10 mg/dL and abnormal kappa/lambda ratio

PRIOR/CONCURRENT THERAPY:

* No anti-myeloma treatments within 14 days before the start of study treatment.
* Must have recovered from side effects of prior treatments.

PATIENT CHARACTERISTICS:

Performance Status

• ECOG 0, 1, or 2

Bone Marrow Reserve

* Absolute neutrophil count (AGC/ANC) ≥ 1000/uL
* Platelets ≥ 30,000/uL
* Hemoglobin ≥ 8g/dL
* Absolute lymphocytes ≥ 800/uL
* Leukocytes ≥ 3,000/uL

Renal Function

• Glomerular Filtration Rate (GFR) > 40mL/min or Serum creatinine ≤ 1.5 X ULN

Hepatic Function

* Total bilirubin ≤ 2.0 X ULN
* AST, ALT, ALP ≤ 3.0 X ULN, or ≤ 5.0 X ULN (if liver metastases exist)
* No positive Hep C serology or active Hep B infection

Cardiovascular

* No congestive heart failure < 6 months
* No unstable angina pectoris < 6 months
* No myocardial infarction < 6 months
* No history of ventricular arrhythmias
* No history of supraventricular arrhythmias
* No NYHA Class > II CHF
* No marked baseline prolongation of QT/QTc interval

Pulmonary

• Normal clinical assessment of pulmonary function

Other

* Negative serum pregnancy test if female and of childbearing potential
* Women who are not pregnant or nursing
* Subjects, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* No known autoimmune disease other than corrected hypothyroidism
* No known prior organ allograft or allogeneic transplantation
* Not HIV positive
* No history or evidence of uncontrollable CNS disease
* No psychiatric illness/social situation
* No other illness that in the opinion of the investigator would exclude the subject from participating in the study
* Must provide informed consent and HIPPA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations
* No active systemic infection requiring parenteral antibiotic therapy
* No on-going chronic systemic corticosteroid (>10 mg daily prednisone equivalent) use or other immunosuppressive therapy (a history of mild asthma not requiring therapy is eligible). Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hing C Wong, PhD, Study Chair — Altor BioScience
Locations (4):
- United States (4):
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study
Groups:
- Cohort 7: N-803 - SQ 20 ug/kg: N-803: Intravenous infusion for cohort 1, 2, 3 and 4; subcutaneous injection for cohort 5, 6 and 7; two 6-week treatment cycles: ALT-803 on Day 1, 8, 15, 22; stable or benefitting patients may receive up to two additional 6-week cycles
Period: Overall Study
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg | Cohort 7: N-803 - SQ 20 ug/kg
Started | 3 | 3 | 3 | 3 | 4 | 3 | 0
Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 3 | 2 | 3 | 2 | 4 | 3 | 0
Not completed — Progressive Disease | 3 | 2 | 2 | 1 | 4 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Groups:
- Cohort 1: ALT-803 - IV 1 ug/kg; Cohort 2: ALT-803 - IV 3 ug/kg; Cohort 3: ALT-803 - IV 6 ug/kg; Cohort 4: ALT-803 - IV 10 ug/kg: ALT-803: Intravenous infusion for cohort 1, 2, 3 and 4; two 6-week treatment cycles: ALT-803 on Day 1, 8, 15, 22; stable or benefitting patients may receive up to two additional 6-week cycles
- Cohort 5: ALT-803 - SQ 10 ug/kg; Cohort 6: ALT-803 - SQ 15 ug/kg; Cohort 7: ALT-803 - SQ 20 ug/kg: ALT-803: subcutaneous injection for cohort 5, 6 and 7; two 6-week treatment cycles: ALT-803 on Day 1, 8, 15, 22; stable or benefitting patients may receive up to two additional 6-week cycles
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALT-803 - IV 1 ug/kg | Cohort 2: ALT-803 - IV 3 ug/kg | Cohort 3: ALT-803 - IV 6 ug/kg | Cohort 4: ALT-803 - IV 10 ug/kg | Cohort 5: ALT-803 - SQ 10 ug/kg | Cohort 6: ALT-803 - SQ 15 ug/kg | Cohort 7: ALT-803 - SQ 20 ug/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 0 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (4.16) | 59.3 (6.66) | 63.7 (6.35) | 61.7 (12.1) | 49.8 (22.63) | 67.0 (5.0) |  | 61.5 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 2 | 0 | 2 | 0 | 9
  Male | 1 | 3 | 0 | 1 | 4 | 1 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  White | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Patients with Relapsed or Refractory Multiple Myeloma [Count of Participants; unit: Participants] | 3 | 3 | 3 | 3 | 4 | 3 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: For phase I - Number of Participants with Treatment Emergent Adverse Events that occur or worsen after the first dose of study treatment.
Time Frame: 24 weeks
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3
Participants | 3 | 3 | 3 | 3 | 4 | 3

2. Primary Outcome: Disease Response Rate of Treated Patients
Description: CR- negative SIFE and UIFE, disappearance of any soft tissue plasmacytomas, and < or = to 5% plasma cells in bone marrow VGPR - either + SIFE and UIFE and - SPEP and UPEP or reduction in serum M-protein > or = to 90% and urine m-protein level <100mg per 24h PR - if measurable serum an urine m-protein them reduction of serum m-protein by >=50% and reduction in 24h urinary m protein by >=90% or to <200mg per 24h if unmeasurable serum and urine m-protein then >= 50% decrease in the difference between involve and uninvolved FLC levels If unmeasurable serum and urine m-protein and serum FLC assay then >= 50% reduction in plasma cells, provide baseline bone marrow plasma cell percentage was >=30% In addition to the above listed criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required PD - defined via International Myeloma Working Group uniform response criteria: disease progression SD - not meeting criteria for CR, VGPR, PR or PD
Time Frame: Starts at Week 11 - 12 and Week 23 - 24
Population: Cohort 5: N-803 - SQ 10 ug/kg - one subject only received 2 doses of study drug. This subject is not evaluable for tumor response assessment.
  Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Participants
  Stable Disease | 0 | 1 | 1 | 1 | 0 | 1
  Progressive Disease | 3 | 2 | 1 | 2 | 2 | 2
  Not available to evaluate | 0 | 0 | 1 | 0 | 1 | 0

3. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Half-life (t½)
Description: Half-life (t½) - The period of time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects. In addition, 6 out of 7 SC patients (Cohorts 5 and 6) had insufficient measurable post-tmax sampling to allow for evaluation of the terminal phase-dependent PK parameters (ie, t½, CL/F, Vz/F, AUC0-168, AUC0-∞).
Measure: Mean (Full Range); unit: Hours
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 0 | 1
Hours | 0.773 [0.734 to 0.826] | 2.41 [2.40 to 2.41] | 2.21 [2.02 to 2.39] | 3.07 [2.33 to 4.14] |  | 35.3 [35.3 to 35.3]

4. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Time of the Observed Maximum Concentration (Tmax)
Description: time of the observed maximum concentration (Tmax)
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3
Hours | 0.583 [0.5 to 0.683] | 0.583 [0.5 to 0.633] | 0.65 [0.633 to 0.717] | 0.667 [0.667 to 2.33] | 33.1 [4.22 to 65.9] | 6.0 [2.0 to 20.3]

5. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Maximum Observed Concentration (Cmax)
Description: maximum observed concentration (Cmax)
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3
ng/mL | 8.45 (1.78) | 42.7 (1.76) | 142 (26.6) | 144 (70.7) | 0.383 (0.111) | 1.69 (1.41)

6. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Area Under the Plasma Concentration Curve
Description: Area under the plasma concentration curve from time 0 through the last measurable concentration (AUC0-t).
  PK samples were obtained from the start of treatment until 72 hours. The AUC0-168 and AUC0-inf were calculated with noncompartmental pharmacokinetic analysis equations.
Time Frame: Samples were collected and the AUC was determined at 24 hours and at time t (last measurable concentration). The AUC was calculated for 168 hours and time to infinity.
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects In addition, 6 out of 7 SC patients (Cohorts 5 and 6) had insufficient measurable post-tmax sampling to allow for evaluation of the terminal phase-dependent PK parameters (ie, t½, CL/F, Vz/F, AUC0-168, AUC0-∞).
Measure: Mean (Full Range); unit: hr x ng/mL
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3
hr x ng/mL
  AUC0-t | 10.5 [7.58 to 13.7] | 129 [105 to 166] | 634 [439 to 845] | 808 [577 to 1200] | 13.6 [6.00 to 21.2] | 60.4 [9.61 to 135]
  AUC0-24: number analyzed (Participants) | 3 | 2 | 2 | 3 | 4 | 3
  AUC0-24 | 10.6 [7.62 to 13.8] | 141 [116 to 166] | 731 [618 to 845] | 811 [577 to 1220] | 5.01 [2.91 to 6.69] | 31.1 [11.7 to 65.5]
  AUC0-168: number analyzed (Participants) | 3 | 2 | 2 | 3 | 0 | 1
  AUC0-168 | 10.6 [7.62 to 13.8] | 141 [116 to 166] | 732 [618 to 846] | 813 [578 to 1220] |  | 31.4 [31.4 to 31.4]
  AUC0-inf: number analyzed (Participants) | 3 | 2 | 2 | 3 | 0 | 1
  AUC0-inf | 10.6 [7.61 to 13.7] | 141 [116 to 166] | 732 [618 to 846] | 814 [578 to 1220] |  | 32.5 [32.5 to 32.5]

7. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Clearance (CL)
Description: Clearance (CL)
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
  Cohorts 1-4 - Clearance (CL)
Measure: Mean (Full Range); unit: mL/hr/kg
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg
Number analyzed (Participants) | 3 | 2 | 2 | 3
mL/hr/kg | 99.9 [72.7 to 131] | 22.0 [18.1 to 25.9] | 8.4 [7.09 to 9.71] | 13.7 [8.20 to 17.3]

8. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Vss Volume of Distribution at Steady State
Description: Vss Volume of distribution at steady state is a ratio of the total amount of drug in the body to the plasma concentration of the drugs such that Vd = amount of drug in body/plasma drug concentration
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Measure: Mean (Full Range); unit: mL/kg
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg
Number analyzed (Participants) | 3 | 2 | 2 | 3
mL/kg | 126 [101 to 159] | 71.8 [65.9 to 77.8] | 34.0 [30.2 to 37.8] | 62.8 [39.0 to 78.0]

9. Secondary Outcome: Immunogenicity - Anti-drug Antibody (ADA)
Description: Number of patients with a positive Anti-drug Antibody (ADA) result
Time Frame: From Baseline up to Week 12
Population: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 2 | 3 | 1 | 2 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Apparent (Extravascular) Clearance (CL/F)
Description: Apparent (Extravascular) Clearance (CL/F)
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: In addition, 6 out of 7 SC patients (Cohorts 5 and 6) had insufficient measurable post-tmax sampling to allow for evaluation of the terminal phase-dependent PK parameters (ie, t½, CL/F, Vz/F, AUC0-168, AUC0-∞).
Measure: Mean (Full Range); unit: mL/hr/kg
Arm/Group | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 0 | 1
mL/hr/kg |  | 462 [462 to 462]

11. Secondary Outcome: Characterization of the Pharmacokinetic Profile - Apparent (Extravascular) Volume of Distribution (Vz/F)
Description: Apparent volume of distribution is a ratio of the total amount of drug in the body to the plasma concentration of the drugs such that Vd = amount of drug in body/plasma drug concentration
Time Frame: PK timepoint up to 72 hours +/- 6 hours
Population: as for outcome 6
Measure: Mean (Full Range); unit: mL/kg
Arm/Group | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg
Number analyzed (Participants) | 0 | 1
mL/kg |  | 23500 [23500 to 23500]

ADVERSE EVENTS:
Time Frame: Treatment-related and non-treatment-related adverse events were monitored/assessed up to 33 weeks. Patients who have an on-going study drug-related SAE upon study completion/discontinuation will be contacted by PI/designee until event is resolved/determined to be irreversible, up to 33 weeks.
Description: Cohort 7: N-803 - SQ 20 ug/kg did not enroll any subjects
Groups:
- Cohort 1: N-803 - IV 1 ug/kg; Cohort 2: N-803 - IV 3 ug/kg; Cohort 3: N-803 - IV 6 ug/kg; Cohort 4: N-803 - IV 10 ug/kg: N-803: Intravenous infusion for cohort 1, 2, 3 and 4; two 6-week treatment cycles: ALT-803 on Day 1, 8, 15, 22; stable or benefitting patients may receive up to two additional 6-week cycles
- Cohort 5: N-803 - SQ 10 ug/kg; Cohort 6: N-803 - SQ 15 ug/kg; Cohort 7: N-803 - SQ 20 ug/kg: N-803: subcutaneous injection for cohort 5, 6 and 7; two 6-week treatment cycles: ALT-803 on Day 1, 8, 15, 22; stable or benefitting patients may receive up to two additional 6-week cycles
Arm/Group | Cohort 1: N-803 - IV 1 ug/kg | Cohort 2: N-803 - IV 3 ug/kg | Cohort 3: N-803 - IV 6 ug/kg | Cohort 4: N-803 - IV 10 ug/kg | Cohort 5: N-803 - SQ 10 ug/kg | Cohort 6: N-803 - SQ 15 ug/kg | Cohort 7: N-803 - SQ 20 ug/kg
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 1/3 | 0/3 | 3/4 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 0/3 | 3/4 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: N-803 - IV 1 ug/kg (N=3) | Cohort 2: N-803 - IV 3 ug/kg (N=3) | Cohort 3: N-803 - IV 6 ug/kg (N=3) | Cohort 4: N-803 - IV 10 ug/kg (N=3) | Cohort 5: N-803 - SQ 10 ug/kg (N=4) | Cohort 6: N-803 - SQ 15 ug/kg (N=3) | Cohort 7: N-803 - SQ 20 ug/kg (N=0)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: N-803 - IV 1 ug/kg (N=3) | Cohort 2: N-803 - IV 3 ug/kg (N=3) | Cohort 3: N-803 - IV 6 ug/kg (N=3) | Cohort 4: N-803 - IV 10 ug/kg (N=3) | Cohort 5: N-803 - SQ 10 ug/kg (N=4) | Cohort 6: N-803 - SQ 15 ug/kg (N=3) | Cohort 7: N-803 - SQ 20 ug/kg (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Administration site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 3 | 0 | 2 | 1 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 2 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 1 | 2 | 3 | 3 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 0 | 1 | 0 | 0
Haptoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lymphocyte count decreased (Infections and infestations) | 1 | 1 | 0 | 2 | 3 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 2 | 2 | 2 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 2 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 1 | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extradural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT02099539/Prot_SAP_000.pdf